CLINICAL TRIAL: NCT02995174
Title: Will Perceptual Learning Via Video Game Playing Improve Visual Acuity, Stereopsis and Fixation Stability in Mild Amblyopes? Part 2 Study
Brief Title: Will Perceptual Learning Via Video Game Playing Improve Visual Acuity Stereopsis & Fixation Stability in Mild Amblyopes?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Carly Lam, Professor, The Hong Kong Polytechnic University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HMRF11122991
Record Dates: First submitted 2016-12-14; First posted 2016-12-16 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Amblyopia
Keywords: amblyopia; fixation stability; perceptual learning
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (dichoptic video game play) (Experimental): Mild amblyopic subjects will be asked to play dichoptic video game in an i-Pod touch device for 1 hour per day in 6 weeks.
  Interventions: Device: Dichoptic video game in an i-Pod touch device
- Control (video game play) (Placebo Comparator): Mild amblyopic subjects will be asked to play video game in an i-Pod touch device for 1 hour per day in 6 weeks.
  Interventions: Device: Video game in an i-Pod touch device

INTERVENTIONS:
Device: Dichoptic video game in an i-Pod touch device — Amblyope will wear a pair of red green goggles and play the video game with 'contrast-balanced' images displayed on the screen of an i-Pod touch device. The eye with weaker eyesight will see the image with high contrast, and the good eye will see the image with low contrast. The subject will play the game one hour per day for 6 weeks.
  Arms: Intervention (dichoptic video game play)
Device: Video game in an i-Pod touch device — Amblyope will wear a pair of red green goggles and play the video game with equal contrast images displayed on the screen of an i-Pod touch device. Both eyes will see the image of same contrast. The subject will play the game one hour per day for 6 weeks.
  Arms: Control (video game play)

SUMMARY:
Contrast balanced dichoptic videogame training has been found to improve sensory functions in adults with amblyopia; best corrected distance visual acuity (BCVA) and stereopsis, but its effect on motor function, namely amblyopic eye fixation stability, is unknown. Furthermore, the effect of treatment in cases of mild amblyopia is not well understood. The aim of this study is to find out the difference on fixation stability, BCVA and stereopsis in mild amblyopes after 6 weeks' contrast balanced dichoptic video game training.

DETAILED DESCRIPTION:
Objectives: To assess the change of fixation stability as well as visual acuity and stereopsis before and after training mild amblyopia by perceptual learning through dichoptic video game playing.

Hypothesis: It has been shown that the visual acuity, stereopsis and fixation stability are compromised in amblyopic eye. Perceptual learning via video game playing has been found effective in improving visual acuity and stereoacuity in moderate and severe amblyopic eyes, but there is no study on such treatment in mild amblyopia. In this study, we hypothesize that fixation stability, visual acuity and stereopsis will be improved after training by dichoptic video game playing in mild amblyopia.

Methods: Participants (aged 7 or above) with Best Corrected Visual Acuity (BCVA) ≤ 0.28 logMAR in the amblyopic eye and an interocular acuity difference ≥ 0.2 logMAR will be recruited. An anaglyphic, contrast balanced dichoptic video game will be provided on an i-Pod Touch (Apple Inc.) for 6 weeks of home-based training (60 mins per day). Fixation stability quantified using bivariate contour ellipse area (BCEA by micro-perimeter (MP) Nidek MP-1), BCVA and stereopsis will be assessed before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Best corrected VA in amblyopic eye ≤ 0.28 log MAR, fellow eye VA with an interocular VA difference ≥ 0.20 log MAR;
* Amblyopia could be in form of strabismic, anisometropic and mixed (both strabismic and anisometropic)
* Able to complete 3 successful measurements (each with 30 seconds fixation) of BCEA by the MP-1 systems in each eye
* Able to align the nonius cross (≤10mm horizontal error and 5mm vertical error) in the i-Pod game

Exclusion Criteria:

* Myopia of spherical equivalent power > -6.0 diopter in either eye
* Previous intraocular surgery
* any types of ocular pathology (e.g. media opacities or retinal lesion)
* Previous or current history of neurological problem

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-08; Primary Completion 2017-12-18 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in fixation stability (in terms of Bivariate contour ellipse area in degree square) in the amblyopic eye after 6 weeks dichoptic video game playing in mild amblyopes | 6 weeks
  Change in fixation stability (in terms of Bivariate contour ellipse area in degree square) in the amblyopic eye after 6 weeks dichoptic video game playing in mild amblyopes. The 95% bivariate contour ellipse area will be adopted in units of degree square.

SECONDARY OUTCOMES:
Change in best corrected visual acuity (in log MAR) in the amblyopic eye after 6 weeks dichoptic video game playing in mild amblyopes | 6 weeks
  Change in best corrected visual acuity (in log MAR) in the amblyopic eye after 6 weeks dichoptic video game playing in mild amblyopes. Best corrected visual acuity will be measured in log MAR unit.
Change in stereopsis (in arc sec) after 6 weeks dichoptic video game playing in mild amblyopes | 6 weeks
  Change in stereopsis (in arc sec) after 6 weeks dichoptic video game playing in mild amblyopes. The Titmus and Randot preschool stereopsis test will be used and the measurements are recorded in ' second of arc'.

CONTACTS AND LOCATIONS:
Overall Officials: Carly Lam, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Birch EE, Li SL, Jost RM, Morale SE, De La Cruz A, Stager D Jr, Dao L, Stager DR Sr. Binocular iPad treatment for amblyopia in preschool children. J AAPOS. 2015 Feb;19(1):6-11. doi: 10.1016/j.jaapos.2014.09.009. PMID 25727578
- [Background] Birch EE, Subramanian V, Weakley DR. Fixation instability in anisometropic children with reduced stereopsis. J AAPOS. 2013 Jun;17(3):287-90. doi: 10.1016/j.jaapos.2013.03.011. PMID 23791411
- [Background] Chung ST, Kumar G, Li RW, Levi DM. Characteristics of fixational eye movements in amblyopia: Limitations on fixation stability and acuity? Vision Res. 2015 Sep;114:87-99. doi: 10.1016/j.visres.2015.01.016. Epub 2015 Feb 7. PMID 25668775
- [Background] Gonzalez EG, Wong AM, Niechwiej-Szwedo E, Tarita-Nistor L, Steinbach MJ. Eye position stability in amblyopia and in normal binocular vision. Invest Ophthalmol Vis Sci. 2012 Aug 9;53(9):5386-94. doi: 10.1167/iovs.12-9941. PMID 22789926
- [Background] Guo CX, Babu RJ, Black JM, Bobier WR, Lam CS, Dai S, Gao TY, Hess RF, Jenkins M, Jiang Y, Kowal L, Parag V, South J, Staffieri SE, Walker N, Wadham A, Thompson B; BRAVO study team. Binocular treatment of amblyopia using videogames (BRAVO): study protocol for a randomised controlled trial. Trials. 2016 Oct 18;17(1):504. doi: 10.1186/s13063-016-1635-3. PMID 27756405
- [Background] Hess RF, Babu RJ, Clavagnier S, Black J, Bobier W, Thompson B. The iPod binocular home-based treatment for amblyopia in adults: efficacy and compliance. Clin Exp Optom. 2014 Sep;97(5):389-98. doi: 10.1111/cxo.12192. Epub 2014 Aug 18. PMID 25131694
- [Background] Li SL, Jost RM, Morale SE, Stager DR, Dao L, Stager D, Birch EE. A binocular iPad treatment for amblyopic children. Eye (Lond). 2014 Oct;28(10):1246-53. doi: 10.1038/eye.2014.165. Epub 2014 Jul 25. PMID 25060850
- [Background] Shaikh AG, Otero-Millan J, Kumar P, Ghasia FF. Abnormal Fixational Eye Movements in Amblyopia. PLoS One. 2016 Mar 1;11(3):e0149953. doi: 10.1371/journal.pone.0149953. eCollection 2016. PMID 26930079
- [Background] Subramanian V, Jost RM, Birch EE. A quantitative study of fixation stability in amblyopia. Invest Ophthalmol Vis Sci. 2013 Mar 19;54(3):1998-2003. doi: 10.1167/iovs.12-11054. PMID 23372053
- [Background] To L, Thompson B, Blum JR, Maehara G, Hess RF, Cooperstock JR. A game platform for treatment of amblyopia. IEEE Trans Neural Syst Rehabil Eng. 2011 Jun;19(3):280-9. doi: 10.1109/TNSRE.2011.2115255. Epub 2011 Feb 17. PMID 21335317